CLINICAL TRIAL: NCT02419664
Title: Ga-68-DOTATOC -PET in the Management of Pituitary Tumours
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The hypothesis we had that we could predict the growth rate from PET uptake could not be confirmer and 3-year follow up was no longer considered motivated
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ga-PET version 8 (141017); 2010-020482-24 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-04-17 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pituitary Tumours
Keywords: pituitary; pituitary adenomas; Ga-PET; Acromegaly; TSHomas; Cushing
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases; Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 DOTATOC PET in pituitary adenomas (Experimental): To give Ga-68 DOTATOC in pituitary patients doing PET/CT
  They are compared with Ga-68 DOTATOC PET performed in another study on patients with no pituitary disease.
  Interventions: Drug: Gallium-68 DOTATOC PET

INTERVENTIONS:
Drug: Gallium-68 DOTATOC PET — The intervention is to administer Ga-68 DOTATOC in pituitary patients doing PET/CT
  Other Names: Ga-PET

SUMMARY:
Title: Gallium (GA) -68-DOTATOC -PET (positron emission tomography) in the management of pituitary tumours Medical product: Ga-68-DOTATOC in PET/computer tomography (CT) Route of administration: Intravenously Diseases of interest: Pituitary tumours Aim: To study the detection of pituitary tumours with Ga-68-DOTATOC -PET (Ga-PET) and to correlate the tracer expression to somatostatin receptor (sst) occurrence Study design: Prospective non-randomised case-control study with open design with GA-PET before and after pituitary surgery in patients with pituitary tumours Study population: patients with acromegaly (n=10), Cushing's' disease of pituitary origin (n=10), TSH (thyreotropin) producing tumours (TSHomas) (n=5) and non-functioning pituitary adenomas (NFPA) (n=20) Number of patients: 45 Inclusion criteria: Adult man or woman (over 18 years) and naïve, unoperated pituitary tumour with growth hormone (GH) or adrenocorticotrophic hormone (ACTH)) or TSH production or NFPA without treatment with somatostatin analogues (SSA) or dopamine agonists.

Exclusion criteria: Patient who may not attend to the protocol according to the investigators opinion. Pregnancy or lactating. Isolated prolactin producing tumours. Overproduction of gonadotropins. Carcinoids ie ectopic corticotrophin realising factor (CRF) production. Known or suspected allergy to the trial product or related products.

Controls: Adult patients with Thyroid associated ophthalmopathy (TAO) before iv steroid infusion (part of another study see this protocol)- Study variables: Tumour detection, Tracer uptake as Standardised uptake value (SUV) max (SUVmax), SUV hotspot and SUV mean in regions of interests (ROIs) Time schedule: Recruitment of patients 2015-2017. Study termination 3 years later

DETAILED DESCRIPTION:
Background The most common cause to pituitary insufficiency is the pituitary adenoma (PA). PA may be divided into hormone producing PAs and non-functioning PAs (NFPA). Normal pituitary tissue, as well as tissues from PAs, expresses somatostatin receptors (sst). Five subtypes of sst receptors has been characterized.

Magnetic resonance tomography (MRI) presents anatomy, while in vivo diagnostics with somatostatin receptor scintigraphy (SRS) or position emission tomography (PET) reflect the functional properties of the tissue. The SRS have earlier been evaluated for diagnostics of pituitary diseases and has low discriminative ability to differ tumor tissue from normal pituitary tissue even though some secretory tumors and NFPA are seen. The superiority of the PET in diagnostics compared to the SRS is based on higher spatial resolution and a higher tumor to background ratio. Therefore it is of large interest to study Gallium 68 DOTATOC (Ga-PET) i small tumours that exhibit sst, such as in the pituitary, where high resolution is essential to discriminate from normal tissue and to evaluated residual tumor tissue postoperatively.

Aim with the project

To evaluate Ga-PET in the management of pituitary tumors and to seek the answer to the following questions:

1. Is the method of value in primary diagnostics in PAs? Does Ga-PET contribute with more functional information than that given from an conventional MRI?
2. Is the method of value in the follow-up, the detection of residual tumor tissue, and increase the possibility to differ scar tissue from true tumor?
3. Can relapses of PA be detected earlier with Ga-PET than with conventional MRI?
4. Are some of the sub-groups easier to detect that others??
5. Can the pathological-anatomical findings and the immunochemical expression of sst be correlated to the PET findings?
6. Can the treatment with somatostatin analogues be designed from the PET investigation and the sst analysis?

Method The aim is to recruit 10 patients with acromegaly (GH-producing PA), 10 patients with Cushing's disease (ACTH-producing PA), 5 patients with TSH-producing PA (TSHoma) and 20 patients with NFPA and to do Ga-PET before and after the pituitary surgery. In the Cushing patients, the TSHomas and in NFPA Ga-PET will also be dome after 3 years postoperatively to detect recurrences. At surgery, pituitary tissue is taken to investigate hormonal expression, sst and for further molecular genetic studies. At all PET occasions blood specimens from the patients are collected for future analyses. They will be kept in a freezer.

If difficulties to separate the Ga-Pet up-take in tumors from normal pituitary tissue the tumor expression may be enhanced by a somatostatin injection before Ga-PET that suppresses normal tissue.

The pituitary PET of pituitary tumours patients will be compared with the pituitary of patients with thyroid associated tumours performing PET according to the similar protocol in Another study

Significance This study is a pilot study. Ga-PET has not been used in pituitary tumors but there is known from studies in patients with gastrointestinal neuroendocrine tumors that the pituitary is seen on GA-PET. This is a "proof of concept". It addresses some of the clinical problems in the management of pituitary tumors. If the questions addressed in this study will be answered in advantage for PET, PET may be a routine investigation and the patients may avoid invasive procedures and repeated MRI. In addition, the patients may have better information regarding cure or not. If not, the treatment may be tailored from the sst receptor expression. This is of great importance for the patients and for the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Naïve, unoperated pituitary tumour with GH or ACTH or TSH production or NFPA without treatment with somatostatin analogues or dopamine agonists.

Exclusion Criteria:

* Patient who may not attend to the protocol according to the investigators opinion.
* Pregnancy or lactating
* Isolated prolactin producing tumours
* Overproduction of gonadotrophins
* Carcinoids ie ectopic CRF production
* Known or suspected allergy to the trial product or related products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
SUV max in GA-68 DOTATOC in pituitary tumours in comparison to normal pituitary | Baseline
  Maximum Standardized Uptake Value
SUV max in GA-68 DOTATOC in pituitary tumours in comparison to normal pituitary | measured at 6 months +/- 2 weeks from baseline
  Maximum Standardized Uptake Value
SUV max in GA-68 DOTATOC in pituitary tumours in comparison to normal pituitary | measured at 36 months +/- 2 weeks from baseline
  Maximum Standardized Uptake Value

SECONDARY OUTCOMES:
Ga-PET uptake in correlation to sst expression in pituitary tumours, measured as SUVmax which is then used to establish statistical relationship with a cell membrane-based sst-immunohistochemistry (IHC) score" | Baseline
Ga-PET uptake in correlation to sst expression in pituitary tumours, measured as SUVmax which is then used to establish statistical relationship with a cell membrane-based sst-immunohistochemistry (IHC) score" | measured at 6 months +/- 2 weeks from baseline
Ga-PET uptake in correlation to sst expression in pituitary tumours, measured as SUVmax which is then used to establish statistical relationship with a cell membrane-based sst-immunohistochemistry (IHC) score" | measured at 36 months +/- 2 weeks from baseline
Adverse event registration in association to Ga-68 PET | Baseline
Adverse event registration in association to Ga-68 PET | measured at 6 months +/- 2 weeks from baseline
Adverse event registration in association to Ga-68 PET | measured at 36 months +/- 2 weeks from baseline
Detection of tumour recurrence with Ga-PET | measured at 6 months +/- 2 weeks from baseline
Detection of tumour recurrence with Ga-PET | measured at 36 months +/- 2 weeks from baseline

OTHER OUTCOMES:
Dynamic measurements of Ga-68 Dotatoc in the pituitary [include the dynamic measure of SUVmax, blood flow, | Baseline
Dynamic measurements of Ga-68 Dotatoc in the pituitary [include the dynamic measure of SUVmax, blood flow, | measured at 6 months +/- 2 weeks from baseline
Dynamic measurements of Ga-68 Dotatoc in the pituitary [include the dynamic measure of SUVmax, blood flow, | measured at 36 months +/- 2 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson Nyström, Ass Prof, Principal Investigator — Center of Endocrinology and Metabolism, Dep of Endorinology, Sahlgrenska University Hospital, Göteborg, Sweden
Locations (1):
- Center of Endocrinology and Metabolism, Sahlgrenska university Hospital, Gothenburg, Sweden